CLINICAL TRIAL: NCT04734886
Title: Exploratory Study on the Effects of Probiotic Supplementation on SARS-CoV-2 Antibody Response in Healthy Adults
Brief Title: The Effect of Probiotic Supplementation on SARS-CoV-2 Antibody Response After COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Collaborators: BioGaia AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: Provid
Record Dates: First submitted 2020-12-10; First posted 2021-02-02 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-09

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L. reuteri DSM 17938 (Active Comparator): Probiotic compound
  Interventions: Dietary Supplement: L. reuteri DSM 17938 + vitamin D
- Placebo (Placebo Comparator): Placebo compound
  Interventions: Dietary Supplement: Placebo + vitamin D

INTERVENTIONS:
Dietary Supplement: L. reuteri DSM 17938 + vitamin D — 1 * 10^8 CFU of L. reuteri DSM 17938 + 10 ug vitamin D3, two capsules per day for 6 months
  Arms: L. reuteri DSM 17938
Dietary Supplement: Placebo + vitamin D — Placebo tablet + 10 ug vitamin D3, Similar in shape and taste to intervention capsules but without the probiotic components, two capsules per day over six weeks
  Arms: Placebo

SUMMARY:
This study will explore how a well-known probiotic strain L. reuteri DSM 17938 impacts SARS-CoV-2 specific antibody response upon and after infection in healthy adults.

DETAILED DESCRIPTION:
After giving their informed consent, the study subjects will complete screening procedures to assess their eligibility for the study (Visit 1). Participants deemed suitable for the study will be randomized into two study arms (placebo, probiotic) before undergoing a baseline visit (Visit 2) before the start of the intervention period. During the 6-month intervention period, the participants will attend study visits at 3 months (Visit 3) into the intervention as well as at the end of intervention (at 6 months, Visit 4). Blood, saliva, and faecal samples will be collected at visits 2-4. In addition to sampling, during the whole intervention period, the participants will fill out a weekly questionnaire in which they are asked to record any possible symptoms of COVID-19. The participants' dietary habits are assessed via a food frequency questionnaire (FFQ) before the start of the intervention period. Also, the participants are asked to maintain their habitual diet and lifestyle as well as not to consume any other probiotic or prebiotic supplements.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Age between 18-60

Exclusion Criteria:

1. Previous diagnosis of COVID-19 (by positive PCR) or previous confirmation of seropositivity to SARS-CoV-2
2. Body Mass Index over 35 or under 16
3. Current diagnosis of cancer or ongoing cancer treatment in the last 12 months
4. Diabetes mellitus
5. Cardiovascular disorder in need of pharmaceutical treatment
6. Chronic kidney disease
7. Chronic lung disease with decreased lung capacity
8. Chronic liver disease with liver cirrhosis
9. Current diagnosis of dementia, severe depression, major psychiatric disorder, or other incapacity for adequate cooperation
10. Chronic neurological/neurodegenerative disease (e.g. Parkinson's disease)
11. Decreased function of the adrenal cortex (e.g. Addison's disease)
12. Autoimmune disease (e.g. rheumatoid arthritis)
13. Chronic pain syndromes (e.g. fibromyalgia)
14. Pregnancy or breast-feeding
15. Immunodeficiency due to disease or ongoing medical treatment
16. Regular intake of anti-inflammatory and/or other immunosuppressive medication within the last 3 months
17. Use of anti-depressants within the last 3 months
18. Antimicrobial treatment within the last 12 weeks before baseline sampling
19. Regular intake of probiotics, as well as nutritional supplements or herb products that might affect intestinal function within the last 4 weeks if the investigator considers that those could affect study outcome
20. Inability to maintain current diet and lifestyle during the study period
21. Alcohol or drug abuse
22. Any clinically significant present or past disease/condition which the investigator considers to possibly interfere with the study outcome or increase the risk for severe form of COVID-19

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 161 (Actual)
Dates: Start 2020-11-27 (Actual); Primary Completion 2021-09-13 (Actual); Study Completion 2021-09-13 (Actual)

PRIMARY OUTCOMES:
SARS-CoV-2 specific antibodies | 3 months (interim analysis) or at 6 months
  Change in SARS-CoV-2 specific IgG/IgM antibodies in serum between the study arms

SECONDARY OUTCOMES:
Maintenance of SARS-CoV-2 seroconversion in seropositive individuals | 3 months + 6 months
  Change in the maintenance of SARS-CoV-2 specific IgG/IgM antibody levels in serum between the study arms
Duration of COVID-19 symptoms measured by a weekly symptom questionnaire | 3 months + 6 months
  Change in duration of COVID-19 related symptoms between the study arms
Severity of COVID-19 symptoms measured by Ordinal Scale for Clinical Improvement (scale 0-7, a lower score corresponds to a better outcome) | 3 months + 6 months
  Change in severity of COVID-19 related symptoms between the study arms
Secretory IgA (sIgA) antibodies | 3 months + 6 months
  Change in sIgA levels in saliva between the study arms
Blood group A antigen antibodies | 3 months + 6 months
  Change in anti-A levels in serum between the study arms
Blood group B antigen antibodies | 3 months + 6 months
  Change in anti-B levels in serum between the study arms
Tn antigen antibodies | 3 months + 6 months
  Change in anti-Tn levels in serum between the study arms
Innate immune system activation | 3 months + 6 months
  Change in high-sensitive C-reactive protein (hs-CRP) levels in plasma between the study groups
Cytokines | 3 months + 6 months
  Change in TNF-a, IFN-y, IL-1B, IL-4, IL-6, IL-8, IL-10 levels in serum between the study groups
Total antibodies | 3 months + 6 months
  Change in total IgG and IgM levels in serum between the study groups
T cell activation | 3 months + 6 months
  Change in the proportion of SARS-CoV-2 specific T cells of all T cells in blood between the study arms
B cell activation | 3 months + 6 months
  Change in the proportion of SARS-CoV-2 specific B cells of all B cells in blood between the study arms
Intestinal inflammation | 3 months + 6 months
  Change in faecal calprotectin levels between the study arms
Intestinal barrier function | 3 months + 6 months
  Change in I-FABP levels in plasma between the study arms
Indirect marker of intestinal permeability | 3 months + 6 months
  Change in LBP levels in plasma between the study arms

OTHER OUTCOMES:
Composition of intestinal microbiota and COVID-19 related symptoms | 3 months + 6 months
  Correlation of intestinal microbiota composition to duration and severity of COVID-19 related symptoms
Composition of intestinal microbiota and SARS-CoV-2 specific antibody | 3 months + 6 months
  Correlation of intestinal microbiota composition to SARS-CoV-2 specific antibody levels in serum
Composition of intestinal microbiota and inflammatory profile | 3 months + 6 months
  Correlation of intestinal microbiota composition to TNF-a, IFN-y, IL-1B, IL-4, IL-6, IL-8, IL-10 levels in serum

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Brummer, MD, PhD, Principal Investigator — Örebro University, Sweden
Locations (1):
- Örebro University, Örebro, Örebro County, Sweden

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared, results will shared only on group-level

REFERENCES:
- [Background] Lehtoranta L, Pitkaranta A, Korpela R. Probiotics in respiratory virus infections. Eur J Clin Microbiol Infect Dis. 2014 Aug;33(8):1289-302. doi: 10.1007/s10096-014-2086-y. Epub 2014 Mar 18. PMID 24638909
- [Background] Zimmermann P, Curtis N. The influence of probiotics on vaccine responses - A systematic review. Vaccine. 2018 Jan 4;36(2):207-213. doi: 10.1016/j.vaccine.2017.08.069. Epub 2017 Sep 18. PMID 28923425